CLINICAL TRIAL: NCT06620718
Title: Evaluation of Pain and Root Migration Distance After Coronectomy Procedure of Impacted Third Molars Based on Age
Brief Title: Evaluation of Root Migration Distance After Coronectomy of Impacted Third Molars
Acronym: NonRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Osman Fatih Arpag, Associate professor, PhD, Mustafa Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022/49
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Impacted Tooth With Abnormal Positioning
Keywords: coronectomy of impacted third molar tooth

STUDY DESIGN:
Intervention Model Description: A total of 78 patients were initially included in the study, but five patients were excluded from the study due to their failure to attend regular follow-up visit, resulting in a final analysis of 73 patients (Figure 1). These patients were divided into two age groups: The first group, consisting of patients aged 18-30, included 17 males and 23 females. The second group, consisting of patients aged 31-55, included 17 males and 16 females.
Masking Description: measurement the distance of root migration at sixth month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of root migration at sixth month after coronectomy (Other): Seventy three patients were divided into two age groups: The first group, consisting of patients aged 18-30, included 17 males and 23 females. The second group, consisting of patients aged 31-55, included 17 males and 16 females
  Interventions: Procedure: coronectomy

INTERVENTIONS:
Procedure: coronectomy — The inferior alveolar nerve and buccal nerve were blocked with maxicaine anaesthetic solution (articaine hydrochloride 40 mg, epinephrine hydrochloride 0.006 mg). Incisions were applied uniformly across all patients, and a triangular flap technique was employed. After elevating the flap and exposing the bone, the bone overlying the crown of the tooth was removed using a bone round bur to fully visualize the tooth's crown. Once the crown was fully exposed, the crown preparation was initiated at the enamel-dentin junction using a fissure bur. The crown preparation was completed without leaving any sharp edges, and the crown was extracted. Then, the exposed pulp was washed with sterile serum without any further intervention. The surgical area was sutured using 5/0 silk. Analgesic (25 mg of dexketoprofen trometamol twice a day) and antibiotic (125 mg clavulanic acid, 875 mg amoxicilin twice a day) drugs were described.

SUMMARY:
The aims of this study were to investigate postoperative pain, edema, and trismus after coronectomy procedure, to assess the risk of endodontic lesion formation at sixth month, and to determine relationship of the root migration distance with age.

DETAILED DESCRIPTION:
The roots of impacted lower third molars may be associated with the inferior alveolar nerve (IAN). To mitigate this risk and reduce trauma to the patient, a conservative approach involving the removal of the problematic crown portion and leaving the root may be adopted.

This clinical study was conducted between 2021-2022 years and was accordance with the Helsinki Declaration of 1975, as revised 2013. All subjects were informed about the study and clinical procedures and provided written consent The study included 73 patients aged between 18-55 years. These patients were divided into two age groups: The first group, consisting of patients aged 18-30. The second group, consisting of patients aged 31-55.

The coronectomy was surgically performed. Postoperative pain, swelling, and interincisal distance were evaluated based on age. Pain was assessed using a 10 cm Visual Analog Scale (VAS) with patients providing ratings before the operation and on the 3rd and 7th postoperative days. The progresion of endodontic lesion was evaluated in 6 months after coronectomy.

The distance of root migration achieved at 6 months after coronectomy was measured by independent examiner. Calibrated panoramic radiographs were used to determine the level of migration.

The statistical analysis of the data obtained in our study was performed using SPSS software The needed statistical analyses were used for comparison of the data. The Levene test was used for comparison of the root migration distances in the age groups. The significance level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The study focused on applying coronectomy, a more conservative approach, instead of extraction for mandibular third molars associated with the inferior alveolar nerve that were indicated for prosthetic, orthodontic, prophylactic purposes, or those causing pericoronitis

  * Systemically health,
  * To maintain ideal oral hygiene,
  * Absence of caries, pulpal and endodontic lesions in the impacted third molar indicated for extraction
  * No known allergies to any antibiotics, or no use or history of bisphosphonate medication
  * No use of tobacco or any illicit drugs by the patient.
  * Not being pregnant

Exclusion Criteria:

* Other conditions unlike abovementioned items.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
the mesaurement of root migration distance | six months after coronectomy procedure
  the distance from the enamel-cement line of the adjacent tooth to the remaining root or roots after coronectomy.

SECONDARY OUTCOMES:
the percentage of edema | postoperatively 3rd and 7th day after coronectomy
  percentage of edema was measured extraorally
the measurement of the distance of interincisal opening | postoperatively 3rd and 7th day after coronectomy
  maximum interincisal distance was measured using a calliper during the maximum opening of the mouth
the pain assessment | postoperatively 3rd and 7th day after coronectomy
  A 10 cm or 100 mm-Visual Analogue Scale was used for assessment. The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Osman F ARPAĞ, Mr, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashemipour MA, Tahmasbi-Arashlow M, Fahimi-Hanzaei F. Incidence of impacted mandibular and maxillary third molars: a radiographic study in a Southeast Iran population. Med Oral Patol Oral Cir Bucal. 2013 Jan 1;18(1):e140-5. doi: 10.4317/medoral.18028. PMID 23229243
- [Background] Satilmis T, Garip H, Arpaci E, Sener C, Goker K. Assessment of combined local anesthesia and ketamine for pain, swelling, and trismus after surgical extraction of third molars. J Oral Maxillofac Surg. 2009 Jun;67(6):1206-10. doi: 10.1016/j.joms.2008.12.034. PMID 19446205
- [Background] Agbaje JO, Heijsters G, Salem AS, Van Slycke S, Schepers S, Politis C, Vrielinck L. Coronectomy of Deeply Impacted Lower Third Molar: Incidence of Outcomes and Complications after One Year Follow-Up. J Oral Maxillofac Res. 2015 Jun 30;6(2):e1. doi: 10.5037/jomr.2015.6201. eCollection 2015 Apr-Jun. PMID 26229580
- [Background] Ghaeminia H, Meijer GJ, Soehardi A, Borstlap WA, Mulder J, Berge SJ. Position of the impacted third molar in relation to the mandibular canal. Diagnostic accuracy of cone beam computed tomography compared with panoramic radiography. Int J Oral Maxillofac Surg. 2009 Sep;38(9):964-71. doi: 10.1016/j.ijom.2009.06.007. Epub 2009 Jul 28. PMID 19640685
- [Background] Pedersen MH, Bak J, Matzen LH, Hartlev J, Bindslev J, Schou S, Norholt SE. Coronectomy of mandibular third molars: a clinical and radiological study of 231 cases with a mean follow-up period of 5.7years. Int J Oral Maxillofac Surg. 2018 Dec;47(12):1596-1603. doi: 10.1016/j.ijom.2018.06.006. Epub 2018 Jul 14. PMID 30017572
- [Background] Monaco G, de Santis G, Gatto MR, Corinaldesi G, Marchetti C. Coronectomy: a surgical option for impacted third molars in close proximity to the inferior alveolar nerve. J Am Dent Assoc. 2012 Apr;143(4):363-9. doi: 10.14219/jada.archive.2012.0178. PMID 22467696